CLINICAL TRIAL: NCT04256564
Title: Comparison of Two Syringe-free In-plane Techniques in Ultrasound-guided Central Venous Catheterization: Jugular Venous Catheterization With Oblique Approach and Brachiocephalic Catheterization Using Y-shape Image
Brief Title: Comparison of Two Syringe-free In-plane Techniques in Ultrasound-guided Central Venous Catheterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Onur Balaban, MD, MD, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/06OBLVSYSHAPE
Record Dates: First submitted 2020-01-14; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Central Venous Catheter Placement
Keywords: Central venous catheter; Ultrasound; Jugular vein; Brachiocephalic vein; Endocavity micro-convex probe; Y-Shape
MeSH Terms: interventions — Catheterization, Central Venous

STUDY DESIGN:
Intervention Model Description: There will be two parallel groups in each a different central catheterization method will be performed.
Who Masked: Participant
Masking Description: The participant will not be aware of the catheterization technique used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oblique visualization linear probe (Experimental): A linear ultrasound probe will be utilized to place the central catheter into the jugular vein
  Interventions: Procedure: Central venous catheterization
- Y-shape visualization micro-convex probe (Experimental): A micro-convex endocavity ultrasound probe will be utilized to place the central catheter into the brachiocephalic vein
  Interventions: Procedure: Central venous catheterization

INTERVENTIONS:
Procedure: Central venous catheterization — A standard 20 cm (adult-size) 3-port central catheter will be placed to the indicated patients by using standard Seldinger technique (with the assist of a guide wire) under ultrasound guidance

SUMMARY:
Ultrasound guidance has become a standard for central venous catheterization. The aim of this study is to compare jugular venous catheterization by using lateral oblique approach to brachiocephalic catheterization by using Y-shape imaging. The trial is planned as prospective randomized and single-blind study. Eighty patients are planned to include in this study. Patients will be assigned to two groups: Oblique visualization Group (central catheter will be placed to the jugular vein by using ultrasound-guided in-plane syringe-free technique) and Y-shape visualization Group (central catheter will be placed to the brachiocephalic vein by using ultrasound-guided in-plane syringe-free technique). Two groups will be compared in terms of number of puncture attempts, procedural time, time of preprocedural ultrasound scanning, overall success rate, complications, the ease of the catheterization process and ultrasound visibility.

DETAILED DESCRIPTION:
Central venous catheters are frequently placed in the operating rooms, intensive care units and emergency departments for various indications such as intravenous fluid, drug infusion, measurement of cardiac parameters and lack of vascular access. Ultrasound guidance has become a standard for central venous catheterization. The use of ultrasound has reduced the number of puncture attempts, increased success rate and reduced complications. While the central venous catheter is inserted by ultrasound, the vessels and the needle can be imaged in real-time. In plane and out-of-plane imaging techniques can be used during catheterization. The in-plane technique ensures the entire needle visualization in ultrasound images. With the linear ultrasound probe, the vessel and needle are imaged longitudinally in the in-plane technique. When an endocavity (micro-convex) ultrasound probe is used, three central vessels (jugular, subclavian and brachiocephalic veins) are displayed as Y-shape. The advantage of the endocavity (micro-convex) probe is that it can visualize deeper tissues and deep veins, and more tissues can be imaged in wider angle. Both techniques have been successfully applied in central catheter placement. In-plane technique also ensures syringe-free cannulation where blood aspiration with a syringe attached to the needle is not necessary.

The aim of this study is to compare two different ultrasound guided in-plane techniques for central venous catheterization. The investigators planned to compare jugular venous catheterization using a linear probe and lateral oblique approach to brachiocephalic catheterization using a micro-convex probe and Y-shape imaging.

The primary outcomes are number of puncture attempts, success rate at first attempt, overall success rate, procedure time, ultrasound scanning time and rate of complications. Secondary outcomes are visibility of the veins and the needle in ultrasound images.

The trial is a comparison of two different interventional technique and planned as prospective randomized and single-blind study. Patients aged between 18-85 years that are planned central venous catheter placement will be included in the study. Patients included in the study will be assigned into two groups by computer-assisted randomization. In the first group (Oblique visualization Group), central catheter will be placed to the jugular vein by using ultrasound-guided in-plane syringe-free technique. In the second group (Y-shape visualization Group), central catheter will be placed to the brachiocephalic vein by using ultrasound-guided in-plane syringe-free technique Linear ultrasound probe will be used in the first group, and endocavity (micro-convex) ultrasound probe will be used in the second group.

In both groups, the number of puncture attempts, the number of needle redirections, and the procedure time will be recorded. The time of preprocedural ultrasound scanning will be recorded in both groups. In addition, complications during the procedure such as bleeding, hemothorax, pneumothorax, hematoma and carotid vascular injury will be recorded. Overall success rates will be assessed in each group at the end of the study. A catheterization procedure will be considered as "unsuccessful" after third puncture attempt or more than 10 needle redirections are needed or requires a procedure time more than 3 minutes. At this moment, the catheter will be placed to a different region or the investigators will switch to a different approach. The ease of the catheterization process will be scored between 0 and 10 by the investigator performing the process (0: the hardest, 10: the easiest). The ultrasound visibility of the needle, vessels, guide wire and catheter will be scored between 0 and 4 (4: excellent view, 3: good view, 2: Medium, 1: difficult 0: impossible to image). The recorded data will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are planned a central venous catheter placement

Exclusion Criteria:

* Morbid obese patients (body mass index> 40)
* People with severe coagulopathy
* Severe deformity at the neck
* Skin deformity or infection at catheterization site
* Congenital anomalies of central veins

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of puncture attempts | During the whole cannulation procedure, starting from the 1st minute until the end of the procedure
  Number of needle insertions to the catheterization region for placing a catheter
Cannulation procedural time | From the 1st minute through withdrawal of the needle, up to 3 minutes
  Duration of the whole cannulation procedure
Catheterization procedural time | During the procedure, starting from the 1st minute through placement of the catheter; up to 3 minutes
  Duration of the whole catheterization procedure
Number of needle redirections | During the whole cannulation procedure, starting from the 1st minute through the procedure; assessed up to 3 minutes
  Redirections of the needle towards the vessel
Success rate | Through study completion, an average of 4 months
  Overall success rates of the procedures in each group
Success rate at first attempt | Through study completion, an average of 4 months
  Success rate at first attempt of the procedures in each group
Complications | Through study completion, an average of 4 months
  Rate of complications that occur during catheterization procedure

SECONDARY OUTCOMES:
Vessel visualization | Throughout the procedure; up to 3 minutes
  Visualization of the vessels in dynamic ultrasound images
Needle visualization | Throughout the procedure; up to 3 minutes
  Visualization of the needle in dynamic ultrasound images
Guide-wire visualization | Throughout the procedure; up to 3 minutes
  Visualization of the guide-wire in dynamic ultrasound images
Catheter visualization | At the end of catheterization procedure
  Visualization of the catheter in dynamic ultrasound images
Ease of the catheterization process | Throughout the procedure; up to 3 minutes
  A subjective score assigned by the operator on a scale with a minimum value of 0 and maximum value of 10. Higher scores mean a better outcome.
Ultrasound time | Throughout the pre-procedural ultrasonography; up to 10 minutes
  The duration of pre-procedural ultrasound scanning

CONTACTS AND LOCATIONS:
Overall Officials: Onur Balaban, MD., Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Evliya CelebiHospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schmidt GA, Maizel J, Slama M. Ultrasound-guided central venous access: what's new? Intensive Care Med. 2015 Apr;41(4):705-7. doi: 10.1007/s00134-014-3628-6. Epub 2015 Jan 8. No abstract available. PMID 25567384
- [Background] Baidya DK, Chandralekha, Darlong V, Pandey R, Goswami D, Maitra S. Comparative Sonoanatomy of Classic "Short Axis" Probe Position with a Novel "Medial-oblique" Probe Position for Ultrasound-guided Internal Jugular Vein Cannulation: A Crossover Study. J Emerg Med. 2015 May;48(5):590-6. doi: 10.1016/j.jemermed.2014.07.062. Epub 2015 Jan 24. PMID 25630474
- [Background] Mallin M, Louis H, Madsen T. A novel technique for ultrasound-guided supraclavicular subclavian cannulation. Am J Emerg Med. 2010 Oct;28(8):966-9. doi: 10.1016/j.ajem.2009.07.019. Epub 2010 Jan 28. PMID 20887917
- [Background] Ital I, Balaban O, Aydin T. Old probe, new method: Y-shape visualization of central veins using endocavitary transducer via omoclavicular acoustic window. Am J Emerg Med. 2018 Mar;36(3):511-513. doi: 10.1016/j.ajem.2017.07.096. Epub 2017 Jul 31. No abstract available. PMID 28789889
- [Background] Kim SC, Heinze I, Schmiedel A, Baumgarten G, Knuefermann P, Hoeft A, Weber S. Ultrasound confirmation of central venous catheter position via a right supraclavicular fossa view using a microconvex probe: an observational pilot study. Eur J Anaesthesiol. 2015 Jan;32(1):29-36. doi: 10.1097/EJA.0000000000000042. PMID 24384583
- [Background] Matias F, Semedo E, Carreira C, Pereira P. [Ultrasound-guided central venous catheterization - "Syringe-Free" approach]. Rev Bras Anestesiol. 2017 May-Jun;67(3):314-317. doi: 10.1016/j.bjan.2016.08.005. Epub 2016 Sep 17. Portuguese. PMID 27650385
- [Background] Ince I, Ari MA, Sulak MM, Aksoy M. [Comparison of transverse short-axis classic and oblique long-axis "Syringe-Free" approaches for internal jugular venous catheterization under ultrasound guidance]. Braz J Anesthesiol. 2018 May-Jun;68(3):260-265. doi: 10.1016/j.bjan.2017.12.002. Epub 2018 Feb 23. PMID 29478705